CLINICAL TRIAL: NCT02849028
Title: The Clinical Research on the Relationship Between Circadian Rhythm and Gut Microbiota in TBI Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: xhechun1
Record Dates: First submitted 2016-07-21; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Loss of Consciousness of Unspecified Duration; Cerebral Laceration and Contusion; Traumatic Brain Injury
Keywords: gut microbiota; sleep disorder; gut-brain axis; circadian rhythm; Traumatic Brain Injury
MeSH Terms: conditions — Contusions; Brain Injuries, Traumatic; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- TBI Patients with sleep disorder: All the patients should be diagnosed by polysomnographic (PSG)
  Interventions: Behavioral: sleep disorder
- health people: The people have a normal sleep
  Interventions: Behavioral: sleep disorder

INTERVENTIONS:
Behavioral: sleep disorder — The study is to investigate whether exist the relationship between sleep disorder and circadian rhythm of patients with TBI or not.

SUMMARY:
Microbiome studies may be highlighted as crucial in the development of sleep disorder for TBI patients. The microbiota-gut-brain connection may further provide an opportunity for microbiota manipulation to treat the TBI patients with sleep disorders.This study is to investigate whether exist the relationship between sleep disorder and circadian rhythm of patients with TBI or not and focus the study on the potential of the host-microbiota interaction in regulating sleep disorder.

DETAILED DESCRIPTION:
Neuroscientists are probing the connections between intestinal microbes and brain development. The general scaffolding of the brain-gut-enteric microbiota axis includes the central nervous system (CNS), the neuroendocrine and neuroimmune systems, the sympathetic and parasympathetic arms of the autonomic nervous system (ANS), the enteric nervous system (ENS), and of course the intestinal microbiota. These components interact to form a complex reflex network with afferent fibers that project to integrative CNS structures and efferent projections to the smooth muscle. Gut microbiota regulates intestinal and extraintestinal homeostasis. Accumulating evidence suggests that the gut microbiota may also regulate brain function and behavior. Results from animal models indicate that disturbances in the composition and functionality of some microbiota members are associated with neurophysiological disorders, strengthening the idea of a microbiota-gut-brain axis and the role of microbiota as a "peacekeeper" in the brain health. It is now clear that the gut-brain communication is bidirectional. On one hand, changes in the microbial community affect behavior. On the other hand, perturbations in behavior alter the composition of the gut microbiota. Since changes in the composition of the gut microbiota are associated with the behavioral and cognitive alterations, a healthy microbiota community is essential for a normal regulation of the microbiota-gut-brain axis. Among the potential factors regulating the axis, microbial metabolites may be the major mediators.

Seven million traumatic brain injuries (TBIs) occur each year in the many countries. One of the most common sequelae in patients exposed to TBI is disrupted sleep, which is especially common following mild TBI. And another one is intestinal function disorder.

Sleep is governed by the intricate interplay between sleep wake homeostasis and circadian rhythms in the body. These rhythms are largely controlled by the suprachiasmatic nucleus (SCN) of the anterior hypothalamus. Clock genes form the molecular machinery of this circadian system, operating via autoregulatory feedback loops.

Among the vertebrate peripheral tissues that express circadian rhythms is the gastrointestinal system, which exhibit circadian rhythms in gene expression (including clock genes), motility and secretion in vivo and in vitro. These rhythms depend upon a patent molecular clock and they are also coordinated by SCN input via the sympathetic nervous system.

The emerging role of the gut microbiome as an important modulator of gastrointestinal function has recently included the role of circadian rhythms. Recent studies have suggested that microbial signaling plays a critical role in homeostatic maintenance of intestinal function along with the host circadian mechanism.

ELIGIBILITY:
Inclusion Criteria:

* The mild TBI (mTBI) patients with sleep disorder (a short loss of consciousness (< 30 min), and/or a short post-traumatic amnesia (PTA) (< 24 h), a Glasgow Coma Scale (GCS) score between 13 and 15)

Exclusion Criteria:

* The mild TBI patients without sleep disorder and the moderate and severe TBI patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The number of patients is 21 and the health people is 21.
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the relationship between sleep disorder and circadian rhythm of patients with TBI | From two weeks to three months after traumatic brain injury
  use real-time PCR and western blot to examine the mRNA and protein expression of circadian genes, BMAL1, Per2, Cry1, Melatonin, and compare with healthy control individuals.

SECONDARY OUTCOMES:
the relationship between gut microbiota and circadian rhythm of patients with TBI | From two weeks to three months after traumatic brain injury
  the relationship between gut microbiota and circadian rhythm of patients with TBI

CONTACTS AND LOCATIONS:
Overall Officials: Xia Hechun, Bachelor, Study Director — The General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No